CLINICAL TRIAL: NCT05356546
Title: TYRX™ Pocket Health Study
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT21029
Record Dates: First submitted 2022-04-14; First posted 2022-05-02 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Cardiac Disease; Healing Surgical Wounds
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tissue samples at least 2 to 3 centimeters (cm) in diameter will be sampled from the device capsule surrounding the implanted CIED for morphometric and histopathology analysis. Samples may be stored for as long as they may be beneficial for study-related analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants with a previous TYRX™ Absorbable Antibacterial Envelope implant: Participants who previously underwent a transvenous CIED implantation with the market released TYRX™ Absorbable Antibacterial Envelope, used for approved indications per country/region, and are returning for a CIED replacement procedure at least 12 months from the prior CIED implantation will be evaluated in this study.
  Interventions: Other: Study-required procedures include: tissue collection from device capsule, questionnaire collection, and photo collection

INTERVENTIONS:
Other: Study-required procedures include: tissue collection from device capsule, questionnaire collection, and photo collection — Enrolled participants will have already received the TYRX™ Absorbable Antibacterial Envelope and will be clinically indicated to have a replacement with any market-released, commercially available (in the geographies they are used) CIED and lead(s) with or without the use TYRX™ Absorbable Antibacterial Envelope, as prescribed by and used on-label by their physician.

SUMMARY:
Medtronic, Inc. is sponsoring the TYRX™ Pocket Health Study to evaluate the histological and morphometric parameters of the device capsule in participants who underwent a cardiovascular implantable electronic device (CIED) procedure with a TYRX™ Absorbable Antibacterial Envelope and are returning for a CIED replacement procedure.

DETAILED DESCRIPTION:
The TYRX™ Pocket Health Study is a prospective, multi-center, single arm, post-market non-interventional study. This global study is planned to be conducted in geographies including, but not limited to, the United States (US), Canada, and Europe, at approximately 5 to 10 centers and will enroll up to 35 subjects with analyzable tissue samples. All enrolled subjects must have an existing CIED (implantable pulse generator (IPG), cardiac resynchronization therapy pacemaker (CRT-P), implantable cardioverter-defibrillator (ICD) or cardiac resynchronization therapy defibrillator (CRT-D)) that was implanted with the TYRX™ Absorbable Antibacterial Envelope and are returning for a clinically indicated CIED generator replacement without the planned addition of new or revision of existing leads.

ELIGIBILITY:
Inclusion Criteria:

1. Previously underwent a transvenous CIED implantation utilizing TYRX™ Absorbable Antibacterial Envelope and is returning for a CIED replacement procedure without planned addition of new or revision of existing leads at least 12 months from the prior CIED implant with use of TYRX™ Absorbable Antibacterial envelope (TYRX procedure of interest)

   a. Participants with history of one or two prior CIED implantation(s) at current implant site can be included, provided there was no invasive intervention to the pocket since the TYRX procedure of interest, defined by Exclusion Criteria #2
2. Age is ≥ 18 years (or meets age requirements per local law) at time of enrollment
3. Procedure information from participant's TYRX procedure of interest can be obtained

   1. Date of the TYRX procedure of interest
   2. Received a TYRX™ Absorbable Antibacterial Envelope during TYRX procedure of interest
4. Provides signed and dated authorization and/or consent per institution and local requirements
5. Willing and able to comply with the protocol

Exclusion Criteria:

1. Active infection involving the CIED implant site (physical, clinical, or laboratory signs/symptoms consistent with an active infection at time of replacement procedure, including but not limited to pneumonia, urinary tract, cellulitis, endocarditis, or bacteremia)
2. Prior history of requiring invasive intervention to the pocket since the TYRX procedure of interest, including but not limited to lead revisions or CIED infection
3. Prior history of skin infection at CIED implant site since the TYRX procedure of interest
4. Returning for a CIED extraction, system upgrade, CIED replacement with planned lead addition and/or revision, planned lead revision, or pocket revision (e.g., pocket revision due to pain)
5. Currently has or requires a submuscular or right-sided CIED implantation, or a subcutaneous implantable cardioverter defibrillator (S-ICD)
6. Existing Ventricular Assist Device (VAD)
7. Currently receiving hemodialysis or peritoneal dialysis therapy
8. Current therapy with chronic oral immunosuppressive agents or ≥ 20mg/day of Prednisone (or equivalent)
9. Has medical condition or history that precludes participant from participation in the opinion of the Investigator (e.g., too superficial positioning of the CIED)
10. Pregnant or breastfeeding participant or participant of childbearing potential and who is not on reliable form of birth regulation method or abstinence
11. Legally incompetent or otherwise vulnerable
12. Participation in another study that may potentially confound the results of this study. Co-enrollment in concurrent trials is only allowed when documented pre-approval is obtained from Medtronic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with one or more prior transvenous CIED implantation at the current implant site utilizing TYRX™ Absorbable Antibacterial Envelope and are returning for a clinically indicated CIED replacement procedure.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2023-07-06 (Actual); Study Completion 2023-07-06 (Actual)

PRIMARY OUTCOMES:
Morphology of device capsule tissue | CIED Replacement Procedure
  Measurement of capsule wall thickness (measured in millimeters, mm) in tissue sample
Histology of device capsule tissue | CIED Replacement Procedure
  Histopathologic examination of tissue sample for extent of fibrosis, inflammation, vascularization, calcification, and adhesions, based on ordinal scoring scale

CONTACTS AND LOCATIONS:
Locations (9):
- United States (6):
  - Clearwater Cardiovascular Consultants, Clearwater, Florida
  - Tallahassee Research Institute, Tallahassee, Florida
  - The Valley Hospital, Ridgewood, New Jersey
  - New York-Presbyterian Hospital/Weill Cornell Medical Center, New York, New York
  - The Stern Cardiovascular Foundation, Germantown, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Institut Universitaire de Cardiologie et de Pneumologie de Québec (IUCPQ), Québec, Canada
- Policlinico Sant Orsola - Malpighi, Bologna, Italy
- Liverpool Heart and Chest Hospital NHS Foundation Trust, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided